CLINICAL TRIAL: NCT00546754
Title: BP-EASE-A 12-Week, Multicenter, Open-Label, Randomized, Controlled Trial To Compare The Effectiveness of Losartan 50 mg/HCTZ 12.5 mg Titrated as Needed to Losartan 100 mg/HCTZ 25 mg or Valsartan 160 mg/HCTZ 25 mg, in Patients With Essential Hypertension Who Have Not Achieved Target Blood Pressure With
Brief Title: BP-EASE -Effectiveness of Losartan 50 mg/Hydrochlorothiazide (HCTZ) 12.5 mg Versus Valsartan 80 mg/HCTZ 12.5 mg Titrated as Needed in Patients With Essential Hypertension Not Controlled on Monotherapy (0954A-333)
Acronym: EASE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0954A-333; MK0954A-333; 2007_031
Record Dates: First submitted 2007-10-17; First posted 2007-10-19 (Estimated); Results first posted 2010-04-13 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2022-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — hydrochlorothiazide, losartan drug combination; Hydrochlorothiazide

ARMS (2):
- 1 (Experimental): Drug Arm
  Interventions: Drug: losartan potassium (+) hydrochlorothiazide
- 2 (Active Comparator): active comparator
  Interventions: Drug: Comparator: Valsartan (+) Hydrochlorothiazide

INTERVENTIONS:
Drug: losartan potassium (+) hydrochlorothiazide — losartan potassium 50 mg/12.5 Hydrochlorothiazide (HCTZ) titrated as needed to losartan potassium 100 mg/25 mg Hydrochlorothiazide
  Arms: 1
Drug: Comparator: Valsartan (+) Hydrochlorothiazide — Valsartan 80 mg/ Hydrochlorothiazide 12.5 mg/day titrated as needed to valsartan 160 mg/25 mg Hydrochlorothiazide
  Arms: 2

SUMMARY:
To evaluate the blood pressure efficacy between losartan and valsartan at equivalent dosage during a 3 months treatment.

ELIGIBILITY:
Inclusion Criteria:

* An Adult Patient 18 to 75 Years Of Age
* Patient with essential hypertension receiving an antihypertensive agent in monotherapy for at least 4 weeks for whom the antihypertensive agent can (and will) be discontinued and whose blood pressure is not controlled:
* Either systolic or diastolic blood pressure > 140/90 mm Hg up to 180/110 mm Hg (inclusive)
* Either systolic or diastolic blood pressure > 130/80 mm Hg up to 160/100 mm Hg (inclusive) for diabetic patients
* Patient is male or a female who is highly unlikely to conceive as she falls into one of the categories listed below:

  * Surgically sterilized female
  * Postmenopausal female > 45 years of age with > 2 years since her last menses
  * Non-sterilized pre-menopausal female who agrees to: (1) use 2 adequate methods of contraception to prevent pregnancy [either 2 barrier methods or a barrier method plus a hormonal method]; or (2) abstain from heterosexual activity throughout the study starting with Visit 1 and for 14 days after the last dose of study medication; or (3) only engage in heterosexual activity with surgically sterilized male partner(s) throughout the study starting with Visit 1 and for 14 days after the last dose of study medication
  * Patient judged to be in otherwise good, stable health on the basis of medical history and physical examination

Exclusion Criteria:

* Known secondary hypertension of any aetiology (e.g., uncorrected renal artery stenosis, malignant hypertension, or hypertensive encephalopathy)
* Patient Needing An Initiation Of A Lipid Lowering Agent Or A Modification Of His Lipid Therapy At Visit 1 Or During The Study Period (12 Weeks)
* Patient taking allopurinol
* Patient Previously Shown To Be Intolerant To Any Component Of Losartan Valsartan, Or HCTZ Or With A Documented History Of Angioedema/Anaphylaxis
* Patient With Confirmed Clinically Significant Renal Or Hepatic Dysfunction And/Or Electrolyte Imbalance Laboratory Test Within The Last 3 Months Prior To Visit 1: Serum Creatinine > 130 Umol/L Or Creatinine Clearance < 45 Ml/Min, Aspartate transaminase (AST) > 2 Times Above The Normal Range, Alanine transaminase (ALT) > 2 Times Above The Normal Range, Serum Potassium < 3.5 Or > 5.5 Meq/L
* Patient with osteoarthritis who has undergone hip or knee replacement within the last 4 months
* Patient with chronic inflammatory conditions such as rheumatoid arthritis, lupus, inflammatory bowel disease and those that need a chronic inflammatory therapy such as prednisone or other steroid agents
* Patient with symptomatic heart failure (classes 3 and 4)
* Patient with a history of stroke within the last 6 months
* Patient with coronary heart disease: has undergone percutaneous coronary angioplasty, has had coronary artery bypass, has had past myocardial infarction, all that occurred less than 6 months prior to visit 1 or has unstable angina
* Patient having participated in an investigational drug program in the last 30 days (prior to Visit 1)
* Unable or unwilling to comply with the protocol, therefore likely to leave the trial before its completion
* Patient intends to move or to vacation away from home during the course of the study which would interfere with the scheduled visits.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 808 (Actual)
Dates: Start 2007-05-01 (Actual); Primary Completion 2009-04-01 (Actual); Study Completion 2009-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient in: MAY-04-2007
  Last patient out: APRIL-16-2009
  Total number of sites: 163 sites in Canada
Groups:
- Losartan 50 mg/HCTZ 12.5 mg: Patients could be titrated up from losartan 50 mg/hydrochlorothiazide (HCTZ) 12.5 mg to losartan 100 mg/HCTZ 25 mg only if needed to achieve target blood pressure.
- Valsartan 80 mg/HCTZ 12.5 mg: Patients could be titrated up from valsartan 80 mg/HCTZ 12.5 mg to valsartan 160 mg/HCTZ 25 mg only if needed to achieve target blood pressure.
Period: Overall Study
Arm/Group | Losartan 50 mg/HCTZ 12.5 mg | Valsartan 80 mg/HCTZ 12.5 mg
Started | 425 (Number of patients enrolled and randomized) | 383 (Number of patients enrolled and randomized)
Treated | 416 (Patients that received at least one dose of study medication and had 1 follow-up visit) | 373 (Patients that received at least one dose of study medication and had 1 follow-up visit)
Week 6 | 396 | 347
Week 12 | 375 | 334
Completed | 375 | 334
Not Completed | 50 | 49
Not completed — Serious Adverse Event | 1 | 1
Not completed — Adverse Event | 11 | 16
Not completed — Lack of Efficacy | 1 | 1
Not completed — Lost to Follow-up | 9 | 15
Not completed — Protocol Violation | 3 | 0
Not completed — Withdrawal by Subject | 6 | 7
Not completed — Dyspnea | 1 | 0
Not completed — Per Data Query, Less Than 4 Wks Coversyl | 1 | 0
Not completed — Hip Replacement | 1 | 0
Not completed — Suicide | 1 | 0
Not completed — Missing Cooperation | 1 | 0
Not completed — Elevated Creatinine and Potassium levels | 0 | 1
Not completed — Patient's Decision | 0 | 1
Not completed — Missing | 14 | 7

BASELINE CHARACTERISTICS:
Groups:
- Losartan 50 mg/HCTZ 12.5 mg: Patients could be titrated up from losartan 50 mg/hydrochlorothiazide (HCTZ) 12.5 mg to losartan 100 mg/HCTZ 25 mg only if needed to achieve target blood pressure.
  416 number of patients that received at least one dose of study medication and had 1 follow-up visit (intent-to-treat population [ITT])
- Valsartan 80 mg/HCTZ 12.5 mg: Patients could be titrated up from valsartan 80 mg/HCTZ 12.5 mg to valsartan 160 mg/HCTZ 25 mg only if needed to achieve target blood pressure.
  373 - number of patients that received at least one dose of study medication and had 1 follow-up visit (intent-to-treat population [ITT])
- Total: Total of all reporting groups
Arm/Group | Losartan 50 mg/HCTZ 12.5 mg | Valsartan 80 mg/HCTZ 12.5 mg | Total
Number analyzed (Participants) | 416 | 373 | 789
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (11.11) | 58.3 (10.26) | 58.5 (10.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 197 | 180 | 377
  Male | 219 | 193 | 412
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 364 | 326 | 690
  Black | 8 | 13 | 21
  Hispanic | 2 | 0 | 2
  Asian | 34 | 29 | 63
  Native | 4 | 4 | 8
  East Indian | 1 | 0 | 1
  From Middle East | 1 | 0 | 1
  Unknown | 2 | 1 | 3

OUTCOME MEASURES:

1. Secondary Outcome: Change in Systolic Blood Pressure From Baseline to Week 6
Time Frame: Baseline and Week 6
Population: 416 and 373 - number of patients that received at least one dose of study medication and had 1 follow-up visit (ITT population). Information available for 392 and 344 patients at week 6 for Losartan 50/HCTZ 12.5mg and Valsartan 80/HCTZ 12.5mg respectively
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Losartan 50 mg/HCTZ 12.5 mg | Valsartan 80 mg/HCTZ 12.5 mg
Number analyzed (Participants) | 392 | 344
mm Hg | -16.7 (14.70) | -18.2 (13.84)
Statistical Analysis 1: Comparison: Losartan 50 mg/HCTZ 12.5 mg vs Valsartan 80 mg/HCTZ 12.5 mg; Test type: Superiority or Other; p = 0.153, ANOVA

2. Secondary Outcome: Change in Diastolic Blood Pressure From Baseline to Week 6
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Losartan 50 mg/HCTZ 12.5 mg | Valsartan 80 mg/HCTZ 12.5 mg
Number analyzed (Participants) | 392 | 344
mm Hg | -8.4 (9.35) | -9.1 (9.16)
Statistical Analysis 1: Comparison: Losartan 50 mg/HCTZ 12.5 mg vs Valsartan 80 mg/HCTZ 12.5 mg; Test type: Superiority or Other; p = 0.343, ANOVA

3. Secondary Outcome: Number of Patients Achieving Target Blood Pressure at Week 6
Description: Number of Patients Achieving Target Blood Pressure (<140/90 mm Hg and <130/80 mm Hg for diabetics) at week 6
Time Frame: Week 6
Population: 416 and 373 - number of patients that received at least one dose of study medication and had 1 follow-up visit (ITT population). Information available for 393 and 345 patients at week 6 for Losartan 50/HCTZ 12.5mg and Valsartan 80/HCTZ 12.5mg respectively
Measure: Number; unit: Patients
Arm/Group | Losartan 50 mg/HCTZ 12.5 mg | Valsartan 80 mg/HCTZ 12.5 mg
Number analyzed (Participants) | 393 | 345
Patients
  Achieved Target Blood Pressure | 253 | 241
  Did Not Achieve Target Blood Pressure | 140 | 104
Statistical Analysis 1: Comparison: Losartan 50 mg/HCTZ 12.5 mg vs Valsartan 80 mg/HCTZ 12.5 mg; Test type: Superiority or Other; p = 0.118, Fisher Exact

4. Primary Outcome: Change in Systolic Blood Pressure From Baseline to Week 12
Time Frame: Baseline and Week 12
Population: 416 and 373 - number of patients that received at least one dose of study medication and had 1 follow-up visit (ITT population). Information available for 371 and 331 patients at week 12 for Losartan 50/HCTZ 12.5mg and Valsartan 80/HCTZ 12.5mg respectively
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Losartan 50 mg/HCTZ 12.5 mg | Valsartan 80 mg/HCTZ 12.5 mg
Number analyzed (Participants) | 371 | 331
mm Hg | -19.9 (13.79) | -20.8 (13.61)
Statistical Analysis 1: Comparison: Losartan 50 mg/HCTZ 12.5 mg vs Valsartan 80 mg/HCTZ 12.5 mg; Test type: Superiority or Other; p = 0.395, ANOVA

5. Secondary Outcome: Number of Patients Achieving Target Blood Pressure at Week 12
Description: Number of Patients Achieving Target Blood Pressure (<140/90 mm Hg and <130/80 mm Hg for diabetics) at week 12
Time Frame: 12 Weeks
Population: 416 and 373 - number of patients that received at least one dose of study medication and had 1 follow-up visit (ITT population). Information available for 372 and 332 patients at week 12 for Losartan 50/HCTZ 12.5mg and Valsartan 80/HCTZ 12.5mg respectively
Measure: Number; unit: Patients
Arm/Group | Losartan 50 mg/HCTZ 12.5 mg | Valsartan 80 mg/HCTZ 12.5 mg
Number analyzed (Participants) | 372 | 332
Patients
  Achieved Target Blood Pressure | 278 | 253
  Did Not Achieve Target Blood Pressure | 94 | 79
Statistical Analysis 1: Comparison: Losartan 50 mg/HCTZ 12.5 mg vs Valsartan 80 mg/HCTZ 12.5 mg; Test type: Superiority or Other; p = 0.662, Fisher Exact

6. Secondary Outcome: Time to Achieve Target Blood Pressure
Description: Time to achieve the target blood pressure (<140/90 mmHg and <130/80 mmHg for diabetics)
Time Frame: 12 weeks
Population: 416 and 373 - number of patients that received at least one dose of study medication and had 1 follow-up visit (ITT population). Information available for 406 and 360 patients for Losartan 50/HCTZ 12.5mg and Valsartan 80/HCTZ 12.5mg respectively
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Losartan 50 mg/HCTZ 12.5 mg | Valsartan 80 mg/HCTZ 12.5 mg
Number analyzed (Participants) | 406 | 360
Days | 62.3 (1.44) | 57.3 (1.24)
Statistical Analysis 1: Comparison: Losartan 50 mg/HCTZ 12.5 mg vs Valsartan 80 mg/HCTZ 12.5 mg; Test type: Superiority or Other; p = 0.020, Log Rank

7. Secondary Outcome: Change in Uric Acid From Baseline to Week 6
Time Frame: Baseline and Week 6
Population: 416 and 373 - number of patients that received at least one dose of study medication and had 1 follow-up visit (ITT population). Information available for 298 and 269 patients at week 6 for Losartan 50/HCTZ 12.5mg and Valsartan 80/HCTZ 12.5mg respectively
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Losartan 50 mg/HCTZ 12.5 mg | Valsartan 80 mg/HCTZ 12.5 mg
Number analyzed (Participants) | 298 | 269
umol/L | 0.3 (53.12) | 21.7 (55.09)
Statistical Analysis 1: Comparison: Losartan 50 mg/HCTZ 12.5 mg vs Valsartan 80 mg/HCTZ 12.5 mg; Test type: Superiority or Other; p < 0.001, ANOVA

8. Primary Outcome: Change in Diastolic Blood Pressure From Baseline to Week 12
Time Frame: Baseline and Week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Losartan 50 mg/HCTZ 12.5 mg | Valsartan 80 mg/HCTZ 12.5 mg
Number analyzed (Participants) | 371 | 331
mm Hg | -10.6 (9.28) | -10.5 (9.58)
Statistical Analysis 1: Comparison: Losartan 50 mg/HCTZ 12.5 mg vs Valsartan 80 mg/HCTZ 12.5 mg; Test type: Superiority or Other; p = 0.935, ANOVA

9. Secondary Outcome: Change in Uric Acid From Baseline to Week 12
Time Frame: Baseline and Week 12
Population: 416 and 373 - number of patients that received at least one dose of study medication and had 1 follow-up visit (ITT population). Information available for 286 and 253 patients at week 12 for Losartan 50/HCTZ 12.5mg and Valsartan 80/HCTZ 12.5mg respectively
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Losartan 50 mg/HCTZ 12.5 mg | Valsartan 80 mg/HCTZ 12.5 mg
Number analyzed (Participants) | 286 | 253
umol/L | -0.4 (57.02) | 29.9 (64.79)
Statistical Analysis 1: Comparison: Losartan 50 mg/HCTZ 12.5 mg vs Valsartan 80 mg/HCTZ 12.5 mg; Test type: Superiority or Other; p < 0.001, ANOVA

10. Secondary Outcome: Change in Serum Highly Sensitive C-reactive Protein From Baseline to Week 6
Time Frame: Baseline and Week 6
Population: 416 and 373 - number of patients that received at least one dose of study medication and had 1 follow-up visit (ITT population). Information available for 304 and 272 patients at week 6 for Losartan 50/HCTZ 12.5mg and Valsartan 80/HCTZ 12.5mg respectively
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Losartan 50 mg/HCTZ 12.5 mg | Valsartan 80 mg/HCTZ 12.5 mg
Number analyzed (Participants) | 304 | 272
mg/L | 0.8 (26.21) | 0.6 (6.60)
Statistical Analysis 1: Comparison: Losartan 50 mg/HCTZ 12.5 mg vs Valsartan 80 mg/HCTZ 12.5 mg; Test type: Superiority or Other; p = 0.899, ANOVA

11. Secondary Outcome: Change in Serum Highly Sensitive C-reactive Protein From Baseline to Week 12
Time Frame: Baseline and Week 12
Population: 416 and 373 - number of patients that received at least one dose of study medication and had 1 follow-up visit (ITT population). Information available for 279 and 255 patients at week 12 for Losartan 50/HCTZ 12.5mg and Valsartan 80/HCTZ 12.5mg respectively
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Losartan 50 mg/HCTZ 12.5 mg | Valsartan 80 mg/HCTZ 12.5 mg
Number analyzed (Participants) | 279 | 255
umol/L | -0.3 (8.05) | 0.5 (7.20)
Statistical Analysis 1: Comparison: Losartan 50 mg/HCTZ 12.5 mg vs Valsartan 80 mg/HCTZ 12.5 mg; Test type: Superiority or Other; p = 0.218, ANOVA

12. Secondary Outcome: Change in Gamma-Glutamyl Transpeptidase (Gamma-GT) From Baseline to Week 6
Time Frame: Baseline and Week 6
Population: 416 and 373 - number of patients that received at least one dose of study medication and had 1 follow-up visit (ITT population). Information available for 300 and 273 patients at week 6 for Losartan 50/HCTZ 12.5mg and Valsartan 80/HCTZ 12.5mg respectively
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Losartan 50 mg/HCTZ 12.5 mg | Valsartan 80 mg/HCTZ 12.5 mg
Number analyzed (Participants) | 300 | 273
IU/L | -1.8 (21.20) | -0.1 (24.71)
Statistical Analysis 1: Comparison: Losartan 50 mg/HCTZ 12.5 mg vs Valsartan 80 mg/HCTZ 12.5 mg; Test type: Superiority or Other; p = 0.386, ANOVA

13. Secondary Outcome: Change in Gamma-Glutamyl Transpeptidase (Gamma-GT) From Baseline to Week 12
Time Frame: Baseline and Week 12
Population: 416 and 373 - number of patients that received at least one dose of study medication and had 1 follow-up visit (ITT population). Information available for 279 and 254 patients at week 12 for Losartan 50/HCTZ 12.5mg and Valsartan 80/HCTZ 12.5mg respectively
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Losartan 50 mg/HCTZ 12.5 mg | Valsartan 80 mg/HCTZ 12.5 mg
Number analyzed (Participants) | 279 | 254
IU/L | -0.7 (21.44) | -0.0 (24.45)
Statistical Analysis 1: Comparison: Losartan 50 mg/HCTZ 12.5 mg vs Valsartan 80 mg/HCTZ 12.5 mg; Test type: Superiority or Other; p = 0.725, ANOVA

ADVERSE EVENTS:
Arm/Group | Losartan 50 mg/HCTZ 12.5 mg | Valsartan 80 mg/HCTZ 12.5 mg
Serious Adverse Events (participants affected / at risk) | 11/425 | 5/383
Other Adverse Events (participants affected / at risk) | 56/425 | 57/383
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Losartan 50 mg/HCTZ 12.5 mg (N=425) | Valsartan 80 mg/HCTZ 12.5 mg (N=383)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Barrett's oesophagus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Critical illness polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 2 (2)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Losartan 50 mg/HCTZ 12.5 mg (N=425) | Valsartan 80 mg/HCTZ 12.5 mg (N=383)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Visual disturbance (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Dyspepsia (General disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomach discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Asthenia (General disorders) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Feeling abnormal (General disorders) | 1 (1) | 0 (0)
Inflammation (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Slugishness (General disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Mastitis (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Back sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incorrect does administered (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Neck injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrong technique in drug usage process (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Blood creatinine increased (Investigations) | 2 (2) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1)
Blood potassium abnormal (Investigations) | 0 (0) | 1 (1)
Blood potassium increased (Investigations) | 3 (3) | 1 (1)
Blood pressure decreased (Investigations) | 0 (0) | 1 (1)
C-Reactive protein increased (Investigations) | 7 (7) | 3 (3)
Cardiac murmur (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 4 (4)
Headache (Nervous system disorders) | 4 (4) | 4 (4)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Mood swings (Psychiatric disorders) | 0 (0) | 1 (1)
Renal impairment (Psychiatric disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Inguinal hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.